CLINICAL TRIAL: NCT03695419
Title: Prevalence of New Psychoactive Substances Use Among Outpatient of Addiction Management Clinic in Assiut University Hospital
Brief Title: Prevalence of New Psychoactive Substances Use
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AAEsraa, Princible investigator, Assiut University
Other Study IDs: PONPSUAOOAMCIAUH
Record Dates: First submitted 2018-09-29; First posted 2018-10-04 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the United Nations Office on Drugs and Crime [UNODC] World Drug Report, the annual prevalence of drug use seemed to be stable for the past few years. However, new psychoactive substances (NPS) have increased drastically in both supply and demand.Many NPS were discovered at the same time as other drugs, and it was simply, for whatever reasons, these other drugs became popular. The majority of these substances are chemicals produced by tweaking or altering the molecular structure of previous well-known psychoactive agents such as cannabis, cocaine, methylenedioxymeth-amphetamine (or MDMA, commonly known as ecstasy), and lysergic acid diethylamide (or LSD), which are being sold as "legal highs," "research chemicals," "herbal highs," "party pills," or "plant food" in an attempt to stay ahead of the law prohibiting the sale and use of psychoactive drugs.Substance abuse rates in Egypt have hit 10%, or double the global average. Tramadol is the most abused substance, followed by cannabis and heroin.In the past two years, two new drugs - known as Strox and Voodoo - have hit the Egyptian market.Voodoo is a combination of an aromatic plant, like marjoram or incense, which is infused with a synthetic cannabinoid that is up to 100 times as powerful as natural marijuana. Shabu is another name for methamphetamine hydrochloride, also known as crystal meth. Meth is a highly addictive stimulant that causes its user irreversible harm, physically and mentally. Pregabalin is increasingly being reported as possessing a potential for misuse.

DETAILED DESCRIPTION:
In 2014, the estimated population who were suffering from drug abuse and drug-related disorders reached over 29 million worldwide, making it a global health challenge. Moreover, 43.5 per million people die annually from associated drug use. According to the United Nations Office on Drugs and Crime [UNODC] World Drug Report, the annual prevalence of drug use seemed to be stable for the past few years. However, new psychoactive substances (NPS) have increased drastically in both supply and demand.

The term "new psychoactive substances" had been legally defined earlier by the European Union as a new narcotic or psychotropic drug, in pure form or in a preparation, that is not scheduled under the Single Convention on Narcotic Drugs of 1961 or the Convention on Psychotropic Substances of 1971, but which may pose a public health threat comparable to that posed by substances listed in those conventions. Although the NPS terminology seems to imply the creation of novel drugs, many are not new. In fact, most psychoactive drugs (that later became abused) have been in use for at least a century. Many NPS were discovered at the same time as other drugs, and it was simply, for whatever reasons, these other drugs became popular. The majority of these substances are chemicals produced by tweaking or altering the molecular structure of previous well-known psychoactive agents such as cannabis, cocaine, methylenedioxymeth-amphetamine (or MDMA, commonly known as ecstasy), and lysergic acid diethylamide (or LSD), which are being sold as "legal highs," "research chemicals," "herbal highs," "party pills," or "plant food" in an attempt to stay ahead of the law prohibiting the sale and use of psychoactive drugs.

On the basis of that definition, European Monitoring Centre for Drugs and Drug Addiction (EMCDDA) identified the following groups of substances covered by its early warning system on NPS:

* Phenethylamines, which encompass a wide range of substances that may exhibit stimulant, entactogenic or hallucinogenic effects.
* Tryptamines, which include a number of substances that have predominantly hallucinogenic effects.
* Piperazines, which are represented, inter alia, by mchlorophenylpiperazine (mCPP) and BZP, both of which are central nervous system stimulants.
* Synthetic cathinones, which have stimulant effects. The main cathinone derivatives are the semi-synthetic methcathinone and the synthetic compounds mephedrone, methylone and MDPV.
* Synthetic cannabinoids are functionally similar to THC, the active compound of cannabis.
* Other substances reported to the early warning system include various plant-derived and synthetic psychoactive substances (e.g. indanes, benzodifuranyls, narcotic analgesics, synthetic cocaine derivatives, ketamine and phencyclidine derivatives), which do not strictly belong to any of the above-mentioned drug families. Also included are a number of medicinal products and derivatives.

NPS are formulated in a variety of forms, and when sold in the market, many contain mixtures of different substances some including controlled drugs. Smoked, ingested, snorted, or injected NPS can produce a variety of psychotropic effects, which can be similar to those related to the controlled substances they contain or to the chemical entities that they are derived from. Based on their clinical effects, NPS can be classified as stimulants, empathogens-entactogens, sedative-hypnotic-anxiolytics, dissociatives, and hallucinogens. Alternatively, they can be classified according to their chemical class as phenethylamines, piperazines, tryptamines, synthetic cathinones, alkylindoles (synthetic cannabinoids), and arylcyclohexylamines.

Substance abuse rates in Egypt have hit 10%, or double the global average. Tramadol is the most abused substance, followed by cannabis and heroin. The ancient culture of Egypt includes an equally ancient history of drug and alcohol abuse. Opium and hashish have been used in Egypt for centuries, and recent tests have found cocaine in mummified remains-a discovery that has confounded historians who considered that the coca plant was purely a South American phenomenon until recent times.It was in the 1980s that use of narcotics began to escalate to serious levels. Currently, Egypt is one of Africa's top cultivators of cannabis and opium poppies. The number of hectares discovered that are dedicated to growing addictive substances has been increasing steadily over the last decade. The amount of "bango"-the local name for marijuana-seizures have also been increasing from 60,000 kg per year up to 80,000 kg and above.

In the past two years, two new drugs - known as Strox and Voodoo - have hit the Egyptian market.Voodoo is a combination of an aromatic plant, like marjoram or incense, which is infused with a synthetic cannabinoid that is up to 100 times as powerful as natural marijuana. The most common brand is "Mister Nice Guy", which is sold in a small bag decorated with a smiley emoticon. The bag has a warning that reads "relaxing incense, not edible". Strox is also made with an aromatic plant like marjoram and incense, which is then sprayed with active medical substances used as pain relievers in case of cramps or stomach aches, like atropine, hyoscine and hyoscyamine. These substances can have psychotropic effects when taken in large doses. Usually, these two drugs are mixed with tobacco and then smoked.

Shabu is another name for methamphetamine hydrochloride, also known as crystal meth. Meth is a highly addictive stimulant that causes its user irreversible harm, physically and mentally.it is a white, odorless substance. Typically, you will find it in a crystal formation or crystalline powder. It tends to be bitter in taste. Sometimes, it's combined with caffeine or other chemicals. Furthermore, it can be packaged in the form of a pill for easy measurement and distribution.

Pregabalin is widely used in neurology, psychiatry and primary healthcare. Pregabalin has been identified within the 30 most prescribed medications in the USA in 2011. In Europe, pregabalin is approved for the treatment of epilepsy (partial seizures), neuropathic pain and generalised anxiety disorder. In the USA, although not approved for anxiety, pregabalin is further approved for fibromyalgia and post-herpetic neuralgia. The molecule is however also often prescribed off-label for a range of clinical conditions, including: bipolar disorder; alcohol/narcotic withdrawal states; attention-deficit/hyperactivity disorder; restless legs' syndrome; trigeminal neuralgia and non-neuropathic pain disorders .Pregabalin is increasingly being reported as possessing a potential for misuse [10]. In the UK, for example, pregabalin prescribing has increased, respectively, by 350 and 150 % in just 5 years. In Norway, Persheim et al. analysed changes for the period 2008-2011 in the drug reimbursement system relating to expenditures for potentially addictive drugs in patients with severe/non-malignant chronic pain, and found that about one-third of the approved applications were for pregabalin. In parallel with this, there is an anecdotally growing black market, with pregabalin being allegedly available without prescriptions through online pharmacies.

Medications obtained by patients for treatment of common ailments, without a prescription from a physician, are known as over-the-counter (OTC) or non-prescription medications. OTC medications provide prevention and treatment for a wide range of conditions, including but not limited to headaches, common cold, musculoskeletal pain, allergies, tobacco dependence, and heartburn. Multiple OTC medications have abuse potential. Commonly abused medications include antihistamines, sleep aids, caffeine, ephedrine, pseudoephedrine, antitussives and expectorants, dextromethorphan, laxatives, anabolic steroids, and sildenafil. Laxatives are abused for weight loss and high antihistamines doses are used for euphoria.

Tropicamide is an antimuscarinic ophthalmic solution used to produce short-acting mydriasis and cycloplegia. Topical abuse of ophthalmic solutions has been reported, but intravenous (IV) abuse of tropicamide seems to be a new phenomenon.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as substance dependence according to DSM-5 criteria.
2. Aged between 18-60 years of both sex.
3. Acceptance to participate in the study.

Exclusion Criteria:

1. Chronic general medical conditions.
2. Patients refused to participate at study
3. History or current bipolar or psychotic disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study group comprised of Egyptians participants. Their age ranged between 18-60 years old, and both men and women are included. They fulfilled the criteria for substance abuse according to DSM-5 criteria. They were selected from the outpatient of addiction management clinic (either admitted to addiction management unit or not) of psychiatric unit of neurology and psychiatry department at Assiut university hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
the prevalence of new psychoactive substance abuse among outpatient of addiction management clinic and patients admitted to addiction management unit of neurology and psychiatry department at Assiut university hospital. | 2years
  All participant will subjected to the following:
  Special sheet designed for the study in department of neurology and psychiatry at Assiut University hospital asking about spychoactive substance use regarding to type, amount, duration,cause of use, and cause for stoppage.
  Addiction severity index Urinary drug screen

CONTACTS AND LOCATIONS:
Overall Officials: Romany H Gabrah, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bozkurt M, Karabulut V, Evren C, Seker M, Kan H. Intravenous Abuse of Tropicamide in Opioid Use Disorder: Presentation of 2 Cases. Subst Abus. 2015;36(2):170-3. doi: 10.1080/08897077.2014.924465. Epub 2014 Jun 3. PMID 24892477